CLINICAL TRIAL: NCT05200949
Title: IMPACT OF SURGICAL EXPERIENCE ON RENAL TRANSPLANT COMPLICATIONS
Brief Title: SURGICAL EXPERIENCE ON RENAL TRANSPLANT COMPLICATIONS
Acronym: IMPACT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 22Uro01
Record Dates: First submitted 2022-01-07; First posted 2022-01-21 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Kidney Transplant Failure
Keywords: Transplant; Kidney
MeSH Terms: interventions — Kidney Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Kidney transplant — Transplant surgery of Kidney

SUMMARY:
Kidney transplantation (KT) failure could be due to surgery dependent factors and particularly surgeon's experience.

Objective: To assess the impact of the surgeon's experience on the post-operative outcomes to know if it safe for young surgeons to perform it.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent Kidney Transplant in CHU of Nice
* Patient for whom a minimum of 12 months follow up is possible.

Exclusion Criteria:

- Patients who underwent a dual Kidney Transplant or a multi-organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patient who was treated with a kidney transplantation in CHU of Nice
Sampling Method: Non-Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Complication post surgery | 1 month after transplant
  complication occurrence using the Clavien Dindo score

SECONDARY OUTCOMES:
function of the transplanted kidney | within 1 year after surgery
  concentration of the creatininemia

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, France

IPD SHARING:
Plan to Share IPD: No
No sharing data plan was established.